CLINICAL TRIAL: NCT00946361
Title: Impaired IGF-1 Generation Causes Protein Catabolism and Poor Growth in Children With Crohn Disease
Brief Title: Impaired Insulin-like Growth Factor-1 (IGF-1) Generation Causes Protein Catabolism and Poor Growth in Children With Crohn Disease
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB09-00036
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2009-07

CONDITIONS: Crohns Disease
MeSH Terms: conditions — Crohn Disease | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic
  Interventions: Other: Examinations

INTERVENTIONS:
Other: Examinations — Growth hormone stimulation testing, Protein turnover, Dexa scan, Bone age x-ray

SUMMARY:
The investigators will prospectively recruit 26 children with moderate - severe active Crohn disease (PCDAI >30). Results will be compared to 26 patients in sustained remission (PCDAI <10 and physician global assessment of remission over the previous 6 months) who are matched for age and gender. Subjects will be studied at baseline and six months. The primary study end-points will be leucine rate of appearance (a measure of protein breakdown) and IGF-1 levels.

This study will test the hypothesis that children with greater disease severity will have worse longitudinal growth and protein catabolism. The investigators will also explore the secondary hypothesis that children with Crohn disease have abnormal IGF-1 generation which is linked to underlying inflammation and disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Crohn disease by endoscopy and histologic samples
* Chronological and/or bone age 6-15 years old
* Tanner 1 - 2
* Willing to participate in our longitudinal evaluation

Exclusion Criteria:

* Concomitant persistent chronic infectious disease
* Inflammatory bowel disease not diagnosed as Crohn disease
* Immunological disorder (excluding Crohn disease)
* Associated severe concomitant chronic illnesses (CF, liver failure)
* Pregnancy

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: GI clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Height velocity | 6 months

SECONDARY OUTCOMES:
Protein catabolism | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dana S Hardin, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital, The Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States